CLINICAL TRIAL: NCT01614054
Title: A Patient-centered Approach to Behavioral Modification in a Tertiary-care University-affiliated Hospital and the Incidence of Smoking Cessation
Brief Title: Nicotine Replacement Provided at a Tertiary Care Hospital
Acronym: N-PATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H12-01080
Record Dates: First submitted 2012-05-28; First posted 2012-06-07 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Nicotine replacement therapy; NRT; Inpatient; General Medicine
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Survey Group (Experimental): Patients will receive a survey along with their meal tray, provided by Food and Nutrition Services. The survey will consist of questions related to smoking habits, desire for NRT and desire for assistance with smoking cessation. The results of these surveys will be collected by allied health professionals and forwarded to the CTU team. The CTU team will then be encouraged to use that information to engage in a discussion with the patient regarding prescription of NRT. It will then be left to the discretion of the HCP whether or not to prescribe NRT taking into account patient preference, absence of contraindications and clinical benefit. All those participating in the survey will be offered referral to a smoking cessation clinic upon discharge.
  Interventions: Other: Survey of patient's smoking habits
- Standard of Care (No Intervention): In the control arm, surveys will also be given out to all patients along with their meal trays. However, these surveys will include only questions related to smoking habits in order to get a baseline number of smokers. The surveys will then be collected by the allied health and nursing staff and forwarded only to the research team. The HCP taking care of the patients will still provide standard of care treatment with NRT and smoking cessation referral as clinically indicated.

INTERVENTIONS:
Other: Survey of patient's smoking habits — Nicotine replacement therapy (inhalers, patches, gum, lozenges) at the discretion of the health care provider
  Arms: Survey Group

SUMMARY:
The purpose of this study is to show that a patient-centered survey asking about smoking habits, with the option for nicotine replacement therapy (NRT) will increase the prescription rates among health care providers (HCP). The investigators also believe that this intervention can also lead to increased referrals to smoking cessation clinics and ultimately increase rates of smoking cessation.

DETAILED DESCRIPTION:
Since the past decade, there has been an increased awareness of the effects of smoking of general health. In 2000, 18.1% of all US deaths were related to tobacco use. Multiple trials have proven that providing nicotine-replacement therapies to help smoking cessation were efficacious with various types of populations. However, smoking has not been eradicated in North America and was associated with a 3.1 million YPLL (years of potential life lost), along with 96.8 billion in productivity losses in the US4.

We are carrying out a study of 200 inpatients on a general medicine ward to attempt to improve prescription rates of nicotine replacement therapy (NRT) and smoking cessation. Our goal is to use a patient centred approach to determine which patients would benefit from NRT and which patients would be in the contemplative stage of smoking cessation. We will want to look at whether a simple, short survey taken by patients can encourage the health care provider (HCP) to provide more NRT and more referrals to a smoking cessation clinic. We hope that this tool will improve the ability of HCP to provide optimal, comprehensive care. The study's findings should help to guide future practices for hospitalized smokers.

Currently, standard treatment involves NRT being prescribed completely at the discretion of the physician. This occasionally involves a discussion with the patient regarding their preferences, but more often is a unilateral decision made by the health care provider. Additionally, we believe that this method misses a lot of potential patients who may benefit from this therapy but are otherwise not identified. We will not be using a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the general medicine ward
* Currently smoking (or quit within the last two weeks)
* 18 years and over
* Able to read in the English language or have a translator present

Exclusion Criteria:

* Non-smokers
* Pregnant or actively trying to conceive
* Recent acute coronary syndrome (within 1 month)
* Active temporo-mandibular joint disease
* Currently on NRT
* Allergy to nicotine
* Acute delirium/chronic dementia
* Inability to complete survey secondary to language/educational issues (if no translator present)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of prescriptions for NRT (as a percentage of the number of active smokers) | 1 month
  By eliciting patient attitudes toward smoking cessation, we aim to increase the rate of prescription of nicotine replacement by 15% on the medical wards at St. Paul's Hospital by 15% over a 1month period.
  We will measure the number of prescriptions for NRT of any kind by referencing pharmacy databases. This will be calculated as a percentage of active smokers.

SECONDARY OUTCOMES:
Number of referrals to a smoking cessation clinic (as a percentage of the number of active smokers) | 1 month
  We hope to increase the number of referrals to smoking cessation clinics by 15% over one month.
  We will measure the number of patients referred for smoking cessation by contacting the clinic and cross-referencing the data by attending physician making the referral. This will be calculated as a percentage of active smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fitzgerald, MD, Principal Investigator — The Lung Centre, University of British Columbia
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada